CLINICAL TRIAL: NCT06823505
Title: Lung Cancer Patients and Parent-child Interaction Experience and Process
Status: Terminated | Type: Observational
Why Stopped: The number of cases received has reached
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202306102RINB
Record Dates: First submitted 2024-06-24; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2023-08

CONDITIONS: Lung Cancer Patients; Parent-child Interaction

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: structured questionnaire — Using the Depression Scale (CES-D), Cancer Self-Efficacy Scale (CASE), Family Peer Relationship Questionnaire (FPRQ), Family Resilience Scale (FRAS) and Parent-Child Relationship Quality Scale

SUMMARY:
Type of study: The goal of this observational study is to explore the relationship between patients with advanced lung cancer and their parent-child interactions during the treatment process, and to understand the impact of the degree of self-differentiation of parents with advanced lung cancer on the physical and mental health of their children. The main questions it aims to answer are:

1. To explore the post-illness adjustment process of patients with advanced lung cancer and the changes in the parent-child relationship among adolescents.
2. To explore the changes in demographic factors-self-belief, mental health, and self-efficacy among patients with advanced lung cancer-and the parent-child relationship among adolescents.
3. Explore the family resilience of patients with advanced lung cancer - family peer relationships, and the interaction between parent-child relationships among adolescents.

DETAILED DESCRIPTION:
This study explores the relationship between late-stage lung cancer patients and their parent-child interactions during the treatment process, and understands the impact of the degree of self-differentiation of parents with late-stage lung cancer on their children's physical and mental health.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced lung cancer aged 40 to 64 years (mid-adulthood).
2. There are lung cancer patients in the family who are teenagers aged 10 to 19 years old.
3. Those who voluntarily participate in this study.
4. Voluntary participants can express themselves orally and in handwriting.

Exclusion Criteria:

1. Single lung cancer patients over 65 years old.
2. Lung cancer patients under 40 years old.
3. Patients diagnosed with early-stage lung cancer.
4. Those who have cognitive impairment and are unable to understand the problem.
5. Those who are unable to express and respond to questions.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with advanced lung cancer aged 40 to 64 years, and have aged 10 to 19 years old teenagers.
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2023-12-17 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Parent-child interaction | one years
  The interaction between patients with advanced lung cancer and their parents and children during the treatment process
Center for Epidemiological Studies Depression Scale | one years
  The CES-D scale is designed to measure an individual's depression level, covering multiple aspects such as depressed mood, guilt, helplessness, decreased appetite, sleep disturbance and psychomotor retardation, with a total of 20 items. The subjects evaluated the frequency of each symptom in the past week using a four-point scale (1 point: never or rarely; 4 points: often). Studies have shown that CES-D has good internal consistency (α=0.85) (Conerly et al., 2002; Given et al., 2004) and reliability (Cronbach's alpha > 0.85) in cancer patients (Hann et al., 2004). al., 1999) , and therefore can effectively assess the level of depression in cancer patients. In short, the CES-D is a validated tool for assessing depression in cancer patients.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei, Taipei City
  - Nation Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No